CLINICAL TRIAL: NCT02262962
Title: Well-Child Care Redesign: A New Model of Care for Children in Low-Income Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Tumaini R Coker, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R40MC21516; K23HD062677 (NIH); R40MC21516 (Other Grant/Funding Number: HRSA)
Record Dates: First submitted 2014-10-03; First posted 2014-10-13 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Preventive Health Services; Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Well-Child Care (No Intervention): No change in Well-Child Visits.
- Redesigned Well-Child Care (Experimental): The Redesigned Well-Child Visits will be enhanced using a newly-designed model of care. Parents will have access to Parent Coach during child's routine well visits, Well Baby Help Line, Well-Visit Planner, and text messaging services (HealthyTxt).
  Interventions: Other: Redesigned Well-Child Care

INTERVENTIONS:
Other: Redesigned Well-Child Care — The Well-Child Visits will be enhanced using a newly-designed model of care. Parents will have access to Parent Coach during child's routine well visits, Well Baby Help Line, Well-Visit Planner, and HealthyTxt Messaging service.
  Arms: Redesigned Well-Child Care

SUMMARY:
The purpose of this research is to design and test a new model for delivery of well-child care (WCC) for children ages 0-3 years in a sample of low-income parents. The investigators used an innovative expert panel and community advisory board process to develop this new model for the delivery of WCC to low-income families in partnership with our partner community pediatric practices. The new model of care utilizes a trained health educator, or "Parent Coach" at every well-visit from 0-3 years of age. The Parent Coach provides a range of services, including health education and guidance, developmental screening, and psychosocial screening and services. The Parent Coach works with the Primary Care Physician to ensure that the family's needs are met for that well-visit. As a part of this new model for well-child care, the parent also uses a web-based tool to help prioritize needs for the visit and complete any necessary pre-visit screening. Parents receive additional education and guidance from a text message service and have access to the Parent Coach outside of the visit.

The randomized controlled trial (RCT) of this new model of care will include 250 families who will be enrolled at participating clinics if the child is under 1 year of age. Parents will receive the intervention for 12 months and will complete surveys to collect data on their experiences of care. Our hypothesis is that this new model of care will be more patient-centered and more effective in providing recommended preventive care services than usual care, and that it will be a sustainable and feasible model for the partner practices.

DETAILED DESCRIPTION:
During Phase 1, we used an innovative expert panel and community advisory board process to develop a new structural model for delivery of well-child care (WCC) to low-income families. The new model of care was developed using a WCC Framework that considered alternative structure for care: non-physician providers (nurses, lay health educators, social workers), non-traditional formats (group visits, internet, phone), and non-clinical locations (daycare centers, home visits, grocery stores) for each of six major WCC visits (physical exam, immunizations/laboratory screening, behavioral/developmental services, anticipatory guidance, psychosocial screenings, and sick visits/after-hours care), as well as a feasible mechanism for provider reimbursement. The model that was developed was a Team-Based Care, Parent Coach Model for WCC.

Recruitment of study participants carried on for approximately six months. We posted flyers in two Los Angeles pediatric clinics. The flyers instructed parents to contact the study investigators by phone or email, or alternatively speak with the office receptionist, if interested in participating. A bilingual (English and Spanish) research associate (RA) was available 2-3 days per week in each clinic site to answer questions that interested parents may have had; that person was also available by phone and email 5 days a week to respond to requests for information. A parent who saw a flyer in the clinic on the day of their visit could have approached the clinic receptionist, expressed an interest in the study, and then directed to either speak with the RA in a private room at the clinic. Additionally, when parents arrived for a visit for a child in the age range specified for the study, they were handed a 1-page flyer regarding the study during check-in at the receptionist's desk. The flyers instructed parents to call, email, or speak in person privately with the study RA if they were interested in participating or needed more information.

Eligible parents were informed of their intervention assignment and were asked for contact information and to complete a 10 minute survey. All parents were informed that they would be contacted 6-months and 12-months post-enrollment to complete two additional surveys. Parents in the intervention group were informed that they may be randomly selected to participate in an additional component to provide study staff with additional information regarding the health services that the parent received during the 12 months that he/she was enrolled in the study.

During enrollment the parents in the intervention group were informed of the additional services available to them. Parents were able to enroll in a text messaging program which provides parents with age-tailored health information through texts. The texts are available in English and Spanish. They contain information such as: car seat safety, dental care for baby and reminders to schedule child's physicals. The second service available to parents is a web-based parent tool called the Well Visit Planner (WVP) tool. The tool gives parents the opportunity to customize their child's upcoming routine physical. The WVP also gives the parents an opportunity to learn about developmental milestones that their child should be meeting. Lastly, parents are given the opportunity to choose priorities to discuss with the physician and the Parent Coach. The data from the pre-visit tool is automatically uploaded to the electronic health record, where red flags indicate areas of further need.

The Parent Coach is also available to intervention patients at the two participating clinics. The Parent Coach is a trained child bilingual health education specialist that will be available at each clinic at least two days a week and over the phone at least one day a week. She is available to help parents schedule appointments and review flagged items on the Well Visit Planner tool. The Parent Coach addresses psychosocial, developmental and behavioral concerns that parents may have. She is also gives parents tips on how parents can help their baby grow and develop. In addition, she is trained to check if the baby is developing normally and if there is reason for concern she will bring it to the attention of the pediatrician at clinic and help parents with referrals for further testing.

Enrollment into the RCT began in June 2013 and ran through December 2013. We enrolled 251 patients over two clinical sites. Half of the participants at each clinic were placed in the control group (n= 125) and the other half in the intervention group (n=126). Research associates are available over the phone and in person at to complete parents follow- up surveys. The 12 month post enrollment surveys are schedule to be completed in December 2014.

ELIGIBILITY:
Inclusion Criteria:

1. Parent or guardian of an infant who is 12 months of age or younger
2. Speaks English or Spanish
3. Is 18 years of age or older

Exclusion Criteria:

1. Has plans to move out of Los Angeles county within the next 12 months
2. Has plans to change the primary care location for the index child within the next 12 months.
3. Parent or guardian is an employee of one of the primary care clinics that are part of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2005-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Receipt of Recommended Preventive Care Services | At 12 months post enrollment
  This is a composite measure

SECONDARY OUTCOMES:
Receipt of Recommended Preventive Care Services | At 6 months post enrollment
  This is a composite measure

CONTACTS AND LOCATIONS:
Overall Officials: Tumaini Coker, MD/MBA, Principal Investigator — UCLA Department of General Pediatrics
Locations (1):
- UCLA Children's Discovery and Innovation Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coker TR, Moreno C, Shekelle PG, Schuster MA, Chung PJ. Well-child care clinical practice redesign for serving low-income children. Pediatrics. 2014 Jul;134(1):e229-39. doi: 10.1542/peds.2013-3775. Epub 2014 Jun 16. PMID 24936004
- [Derived] Coker TR, Chacon S, Elliott MN, Bruno Y, Chavis T, Biely C, Bethell CD, Contreras S, Mimila NA, Mercado J, Chung PJ. A Parent Coach Model for Well-Child Care Among Low-Income Children: A Randomized Controlled Trial. Pediatrics. 2016 Mar;137(3):e20153013. doi: 10.1542/peds.2015-3013. Epub 2016 Feb 10. PMID 26908675